CLINICAL TRIAL: NCT06775548
Title: Effects of Exercises and Vitamins on Oxidative Stress & Inflammatory Markers Among Patients with Depression
Brief Title: Comparing the Effects of Aerobic & Resistance Exercises and Vitamins D & E on Oxidative Stress & Inflammatory Markers Among Patients with Depression
Acronym: TNF; IL-6
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Erum Tanveer, PhD Scholar, Ziauddin University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 86404243ETREH
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Depression Disorders
Keywords: Depression; Oxidative Stress; Inflammatory Markers; Aerobic Exercises; Resistance Exercises; Vitamin E; Vitamin D
MeSH Terms: conditions — Depression | interventions — Exercise; Vitamin E; Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Experimental): Aerobic Exercises with Vitamin E
  Interventions: Other: Aerobic Exercises + Vitamin E
- Group B (Experimental): Resistance Exercises with Vitamin E
  Interventions: Other: Resistance Exercises + Vitamin E
- Group C (Experimental): Aerobic Exercises with Vitamin D
  Interventions: Other: Aerobic Exercises + Vitamin D
- Group D (Experimental): Resistance Exercises with Vitamin D
  Interventions: Other: Resistance Exercises + Vitamin D

INTERVENTIONS:
Other: Aerobic Exercises + Vitamin E — For aerobic exercise, patient will perform cycling. The patient will perform stationary bike with an intensity of 60-85% of MHR by using Karvonean formula for duration of 30 minutes for 4 days/ week. Participants will be advised by the physical therapist to sit on a cycle ergometer with back supported, hands holding the handle bar and feet firmly placed on the pedals.
  The imprint of FITT protcol by ACSM for aerobic exercise will be as follows, Frequency: 4 days/week Intensity: 60-85% of MHR Time: 30 minutes Type: Stationary bike
  Arms: Group A
Other: Resistance Exercises + Vitamin E — The strength training protocol will focus on 10 major muscles of the body. The sessions will be performed for 4 days per week, lasting approximately 30 minutes. The training will be divided in a systematical manner, on first- and third-day participant will perform strength training of upper limb and abdominal muscles that include: Biceps, Triceps, Pectoralis Major, Deltoid, and abdominal muscles. On second and fourth day, participant will perform strength training of lower back and lower limb muscles that include: Latissimus Dorsi, Abdominals, Back Extensors, Hamstrings, Quadriceps and Calf. The intensity of the weight bearing exercises will be calculated using 1 Repetition Maximum (RM) method. The protocol will be divided as follows: 2 days the participant will perform exercises for upper limb and 2 days, patient will perform exercises for lower limb.
  Arms: Group B
Other: Aerobic Exercises + Vitamin D — For aerobic exercise, patient will perform cycling. The patient will perform stationary bike with an intensity of 60-85% of MHR by using Karvonean formula for duration of 30 minutes for 4 days/ week. Participants will be advised by the physical therapist to sit on a cycle ergometer with back supported, hands holding the handle bar and feet firmly placed on the pedals. The imprint of FITT protcol by ACSM for aerobic exercise will be as follows, Frequency: 4 days/week Intensity: 60-85% of MHR Time: 30 minutes Type: Stationary bike
  Arms: Group C
Other: Resistance Exercises + Vitamin D — The strength training protocol will focus on 10 major muscles of the body. The sessions will be performed for 4 days per week, lasting approximately 30 minutes. The training will be divided in a systematical manner, on first- and third-day participant will perform strength training of upper limb and abdominal muscles that include: Biceps, Triceps, Pectoralis Major, Deltoid, and abdominal muscles. On second and fourth day, participant will perform strength training of lower back and lower limb muscles that include: Latissimus Dorsi, Abdominals, Back Extensors, Hamstrings, Quadriceps and Calf. The intensity of the weight bearing exercises will be calculated using 1 Repetition Maximum (RM) method. The protocol will be divided as follows: 2 days the participant will perform exercises for upper limb and 2 days, patient will perform exercises for lower limb.
  Arms: Group D

SUMMARY:
Depression has been ranked as the fourth leading contributor to disability globally. As per data provided by the World Health Organization (WHO), depression affects approximately 3.8% of the global population, constituting approximately 280 million individuals worldwide, with an annual suicide-related mortality of 700,000 people GHDx 2023). Women are 50% more affected with depression as compared to men. Approximately 27.4% have experienced symptoms associated with anxiety and depression in Pakistan. The increasing prevalence and yearly occurrence influenced by the COVID-19 have compelled us to reevaluate the significance of mental well-being. Furthermore, based on the latest data, there has been an increase of 53.2 million cases of depressive disorder worldwide, indicating a growth of 27.6% throughout this pandemic. The prevalence of depression is uniform in both developed and economically challenged nations, independent of cultural background, origin, or ethnicity. Depression has various forms which include major depressive disorder (MDD), bipolar disorder (manic depression), persistent depressive disorder (dysthymia), and seasonal affective disorder (SAD). In the present time, MDD is the leading cause of global disability, contributing to 7.5% of years lived with a disability. (YLD) worldwide, with an estimated annual cost surpassing $US 1 trillion.

The primary etiology of MDD is disturbances in neurotransmitters and neuroendocrine regulation, accompanied by a complex interaction of genetic and environmental factors. In addition to these factors, increasing attention has been directed towards understanding the pathophysiology of MDD through the relationship between oxidative stress and inflammation. Essential enzymatic antioxidants, particularly Glutathione Peroxidase (GPx) and Superoxide Dismutase (SOD), play a crucial role in moderating oxidative stress. Oxidative stress arises from an imbalance between the generation of reactive oxygen species (ROS) and the body's capacity to counteract them. Studies indicate a tendency for reduced GPx and SOD activity in individuals with MDD, leading to heightened oxidative stress.

Furthermore, the involvement of pro-inflammatory cytokines, such as Tumor Necrosis Factor-alpha (TNF) and Interleukin-6 (IL-6), in the inflammatory processes associated with depression is noteworthy. Persistent inflammation is associated with the activation of the kynurenine pathway, triggering the production of neurotoxic metabolites that may contribute to observed neurobiological changes in MDD. Elevated levels of TNF and IL-6, key immune response mediators, are observed in individuals with depression. These cytokines influence neurotransmitter metabolism, disrupt the blood-brain barrier, and activate microglia, spreading neuro-inflammation. The bidirectional interplay between oxidative stress and inflammation establishes a cyclically reinforcing paradigm, amplifying the neurobiological substrates of depression.. Moreover, deficiencies in various vitamins and minerals are significantly associated with Major Depressive Disorder (MDD), including vitamin D and E. Vitamin D and its metabolite calcitriol may act as a defense mechanism for the brain, guarding against the depletion of dopamine and serotonin whereas vitamin E has an antidepressant-like effect.

The management of major depressive disorder encompasses diverse treatment approaches, comprising pharmacological, psychotherapeutic, interventional, and lifestyle modifications, such as incorporating exercise and dietary changes. While the current antidepressants are more effective than placebos in adults with MDD, limitations of antidepressant treatment include a prolonged therapeutic time lag required for the clinical betterment of depressive symptoms and various side effects linked to their usage. These side effects frequently lead to treatment discontinuation by patients. Consequently, adjunctive treatments may play a crucial role in managing this disorder, particularly in cases of treatment resistance.

Engaging in regular exercise exerts a beneficial impact on symptoms commonly associated with depression. The consistent practice of physical activity positively influences various physiological aspects, encompassing neurotransmitter levels, neurotrophic factors, hormonal balance, immune modulation, sleep quality, and cognitive functions. This comprehensive influence collectively provides substantial evidence for the therapeutic effectiveness of exercise in alleviating depressive symptoms. Hence, the objective of the current study is to investigate the outcomes of aerobic and resistance exercises in conjunction with vitamin supplementation on individuals diagnosed with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
A total number of 116 participants will be recruited in the study. After the voluntarily consent, all the participants will be equally divided into four of the treatment group Group-A, B, C and D using envelop method of simple random sampling technique. In addition, a total of 116 sealed envelopes, comprises of 29 envelopes for each group will be presented to the patients. Each patient will be asked to select one envelope of their choice. Upon selection of the envelope, patients will be allocated to the respective group. Thus, each group will comprise of 29 participants Afterwards, pre-assessment will be performed for each patient on all 3 outcome measures i.e. Oxidative stress (SOD & GPX), inflammatory markers (TNF alpha & IL-6) Depression severity (PHQ-9) respectively.

Participants in Group-A will be receiving Aerobic Exercise with Vitamin E, Group-B participants will be receiving Resistance Exercise with Vitamin E, Group C: Aerobic Exercise with Vitamin D, while Group D will be receiving Resistance Exercise with Vitamin D. Whereas, all the groups will be given 48 sessions of their respective protocol, comprising of 30 minutes, 4 times/week for the duration of 12 weeks.

Participants referred to the study will undergo a thorough screening process as discussed below to determine their eligibility.

The recruitment of patients will be conducted by a psychiatrist, adhering to predefined inclusion and exclusion criteria. Patients will undergo screening and be categorized as having Major Depressive Disorder (MDD) if they exhibit at least one of the two primary criteria-depressed mood or anhedonia (the inability to experience pleasure or loss of interest)-along with four or more secondary symptoms persisting for a minimum period of 2 weeks, as per DSM-5 guidelines (American Psychiatric Association, 2013).

They will then be screened through PARQ & YOU questionnaire by physical therapist. Subsequently, the investigator will provide a comprehensive overview of the study to the patients and secure informed consent upon their agreement. Demographic information and pertinent variables, including the duration of the disease and comorbidities, will be documented before the baseline assessment. All patients will adhere to their routine pharmacological care throughout the intervention period.

An orientation session will be arranged before starting the intervention in which the physical therapists in detailed will brief the participants regarding the protocol. The intervention will last for duration of 12 weeks with a total of 48 sessions. First, the participant will perform 1 week of training as part of familiarization phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients with mild to moderate depression, aged between 25-35 years referred by Psychiatrist with no other Psychiatric disease attending the respective unit of Creek General Hospital and Dr. Ziauddin Hospital. (Kivani M et al, 2022, Khan B et al., 2022).
* Individuals both with and without current psychoactive medication (such as antidepressants or anxiolytics) will be enrolled. (O'Sullivan et al., 2023)
* Participants willing to participate to the intervention.

Exclusion Criteria:

* Participants with diagnosed cardiovascular diseases,
* Participants with pregnant women,
* Participants with use of beta-blockers,
* Participants with a history of severe mental illnesses (mentally handicapped),
* Participants with hypertension, hyperparathyroidism,
* Participants with current significant substance or alcohol abuse, ongoing burn-out syndrome, and
* Participants with An elevated suicide risk determined by the Psychiatrist.
* Participants with Prisoners
* Participants with chronic diseases such as liver and renal diseases, mal-absorption syndrome, and other diseases that can affect the level of vitamin D.
* Patients with physical limitations that would prohibit the participation in following exercise protocol.
* Participants consuming dietary supplements two months prior to the intervention.
* Participation in regular exercise during the past 6 months (2 days/week).
* Non cooperative patients and refused to continue the intervention program.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Glutathione Peroxidase and Superoxide Dismutase | Baseline
  Oxidative stress will be assessed in each group using a colorimetric method and commercially available kits. This method involves measuring the optical density at 560 nm of the blue formazan dye produced during the interaction of nitro blue tetrazolium with superoxide radicals generated through the use of xanthine and xanthine oxidase. The Superoxide Dismutase present in the sample works to neutralize the superoxide radicals in the medium, thereby inhibiting the formazan reaction. Specifically, one unit of SOD reduces the nitro blue tetrazolium at a rate of 50% under the specified assay conditions
Glutathione Peroxidase and Superoxide Dismutase | 12 weeks
  Oxidative stress will be assessed in each group using a colorimetric method and commercially available kits. This method involves measuring the optical density at 560 nm of the blue formazan dye produced during the interaction of nitro blue tetrazolium with superoxide radicals generated through the use of xanthine and xanthine oxidase. The Superoxide Dismutase present in the sample works to neutralize the superoxide radicals in the medium, thereby inhibiting the formazan reaction. Specifically, one unit of SOD reduces the nitro blue tetrazolium at a rate of 50% under the specified assay conditions
Inflammatory Markers | Baseline
  TNF and IL-6 will be assessed using commercially available ELISA kits. The procedures for preparing reagents, standards, and serum samples, as well as the overall assay process, will be conducted in accordance with the manufacturer's instructions for each respective ELISA kit. Each ELISA kit plate consisted of 116 microtiter wells, all of which will be coated with antibodies targeting a specific antigenic site of the respective cytokine molecule. The concentrations of IL-6 and TNF will be reported in units of pg/mL and mg/L, respectively
Inflammatory Markers | 12 weeks
  TNF and IL-6 will be assessed using commercially available ELISA kits. The procedures for preparing reagents, standards, and serum samples, as well as the overall assay process, will be conducted in accordance with the manufacturer's instructions for each respective ELISA kit. Each ELISA kit plate consisted of 116 microtiter wells, all of which will be coated with antibodies targeting a specific antigenic site of the respective cytokine molecule. The concentrations of IL-6 and TNF will be reported in units of pg/mL and mg/L, respectively
Patient Health Questionnaire (PHQ-9) | Baseline
  PHQ- 9 is a subjective score for assessing depression severity level. It has 9 questions with a maximum score of 27.
Patient Health Questionnaire (PHQ-9) | 12 weeks
  PHQ- 9 is a subjective score for assessing depression severity level. It has 9 questions with a maximum score of 27.

CONTACTS AND LOCATIONS:
Overall Officials: Erum Tanveer, Principal Investigator — Ziauddin University
Locations (1):
- Ziauddin College of Physical Therapy, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Fu Z, Bo Q, Mao Z, Ma X, Wang C. The reliability and validity of PHQ-9 in patients with major depressive disorder in psychiatric hospital. BMC Psychiatry. 2020 Sep 29;20(1):474. doi: 10.1186/s12888-020-02885-6. PMID 32993604
- [Background] Schuch FB, Deslandes AC, Stubbs B, Gosmann NP, Silva CT, Fleck MP. Neurobiological effects of exercise on major depressive disorder: A systematic review. Neurosci Biobehav Rev. 2016 Feb;61:1-11. doi: 10.1016/j.neubiorev.2015.11.012. Epub 2015 Dec 2. PMID 26657969
- [Background] COVID-19 Mental Disorders Collaborators. Global prevalence and burden of depressive and anxiety disorders in 204 countries and territories in 2020 due to the COVID-19 pandemic. Lancet. 2021 Nov 6;398(10312):1700-1712. doi: 10.1016/S0140-6736(21)02143-7. Epub 2021 Oct 8. PMID 34634250
- [Background] Ross RE, VanDerwerker CJ, Saladin ME, Gregory CM. The role of exercise in the treatment of depression: biological underpinnings and clinical outcomes. Mol Psychiatry. 2023 Jan;28(1):298-328. doi: 10.1038/s41380-022-01819-w. Epub 2022 Oct 17. PMID 36253441
- [Background] Palapar L, Kerse N, Rolleston A, den Elzen WPJ, Gussekloo J, Blom JW, Robinson L, Martin-Ruiz C, Duncan R, Arai Y, Takayama M, Teh R; TULIP Consortium. Anaemia and physical and mental health in the very old: An individual participant data meta-analysis of four longitudinal studies of ageing. Age Ageing. 2021 Jan 8;50(1):113-119. doi: 10.1093/ageing/afaa178. PMID 32939533
- [Background] O'Sullivan D, Gordon BR, Lyons M, Meyer JD, Herring MP. Effects of resistance exercise training on depressive symptoms among young adults: A randomized controlled trial. Psychiatry Res. 2023 Aug;326:115322. doi: 10.1016/j.psychres.2023.115322. Epub 2023 Jun 28. PMID 37429171
- [Background] Nishuty NL, Khandoker MMH, Karmoker JR, Ferdous S, Shahriar M, Qusar MMAS, Islam MS, Kadir MF, Islam MR. Evaluation of Serum Interleukin-6 and C-reactive Protein Levels in Drug-naive Major Depressive Disorder Patients. Cureus. 2019 Jan 11;11(1):e3868. doi: 10.7759/cureus.3868. PMID 30899619
- [Background] Moraes HS, Silveira HS, Oliveira NA, Matta Mello Portugal E, Araujo NB, Vasques PE, Bergland A, Santos TM, Engedal K, Coutinho ES, Schuch FB, Laks J, Deslandes AC. Is Strength Training as Effective as Aerobic Training for Depression in Older Adults? A Randomized Controlled Trial. Neuropsychobiology. 2020;79(2):141-149. doi: 10.1159/000503750. Epub 2019 Oct 28. PMID 31658460
- [Background] Mikola T, Marx W, Lane MM, Hockey M, Loughman A, Rajapolvi S, Rocks T, O'Neil A, Mischoulon D, Valkonen-Korhonen M, Lehto SM, Ruusunen A. The effect of vitamin D supplementation on depressive symptoms in adults: A systematic review and meta-analysis of randomized controlled trials. Crit Rev Food Sci Nutr. 2023 Nov;63(33):11784-11801. doi: 10.1080/10408398.2022.2096560. Epub 2022 Jul 11. PMID 35816192
- [Background] Mandolesi L, Polverino A, Montuori S, Foti F, Ferraioli G, Sorrentino P, Sorrentino G. Effects of Physical Exercise on Cognitive Functioning and Wellbeing: Biological and Psychological Benefits. Front Psychol. 2018 Apr 27;9:509. doi: 10.3389/fpsyg.2018.00509. eCollection 2018. PMID 29755380
- [Background] Maurus I, Hasan A, Roh A, Takahashi S, Rauchmann B, Keeser D, Malchow B, Schmitt A, Falkai P. Neurobiological effects of aerobic exercise, with a focus on patients with schizophrenia. Eur Arch Psychiatry Clin Neurosci. 2019 Aug;269(5):499-515. doi: 10.1007/s00406-019-01025-w. Epub 2019 May 21. PMID 31115660
- [Background] Li J, Wang L, Wang Z, Zhao F, Sun Y, Lu Y, Yang L. Association between suicide attempts and anemia in late-life depression inpatients. BMC Geriatr. 2024 Jan 10;24(1):43. doi: 10.1186/s12877-023-04649-9. PMID 38200429
- [Background] Jamilian M, Shojaei A, Samimi M, Afshar Ebrahimi F, Aghadavod E, Karamali M, Taghizadeh M, Jamilian H, Alaeinasab S, Jafarnejad S, Asemi Z. The effects of omega-3 and vitamin E co-supplementation on parameters of mental health and gene expression related to insulin and inflammation in subjects with polycystic ovary syndrome. J Affect Disord. 2018 Mar 15;229:41-47. doi: 10.1016/j.jad.2017.12.049. Epub 2017 Dec 28. PMID 29306057
- [Background] Imboden C, Gerber M, Beck J, Eckert A, Lejri I, Puhse U, Holsboer-Trachsler E, Hatzinger M. Aerobic Exercise and Stretching as Add-On to Inpatient Treatment for Depression Have No Differential Effects on Stress-Axis Activity, Serum-BDNF, TNF-Alpha and Objective Sleep Measures. Brain Sci. 2021 Mar 24;11(4):411. doi: 10.3390/brainsci11040411. PMID 33805073
- [Background] Nedic Erjavec G, Sagud M, Nikolac Perkovic M, Svob Strac D, Konjevod M, Tudor L, Uzun S, Pivac N. Depression: Biological markers and treatment. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Mar 8;105:110139. doi: 10.1016/j.pnpbp.2020.110139. Epub 2020 Oct 15. PMID 33068682
- [Background] Huang Q, Liu H, Suzuki K, Ma S, Liu C. Linking What We Eat to Our Mood: A Review of Diet, Dietary Antioxidants, and Depression. Antioxidants (Basel). 2019 Sep 5;8(9):376. doi: 10.3390/antiox8090376. PMID 31491962
- [Background] Hidese S, Saito K, Asano S, Kunugi H. Association between iron-deficiency anemia and depression: A web-based Japanese investigation. Psychiatry Clin Neurosci. 2018 Jul;72(7):513-521. doi: 10.1111/pcn.12656. Epub 2018 May 9. PMID 29603506
- [Background] Hasin DS, Sarvet AL, Meyers JL, Saha TD, Ruan WJ, Stohl M, Grant BF. Epidemiology of Adult DSM-5 Major Depressive Disorder and Its Specifiers in the United States. JAMA Psychiatry. 2018 Apr 1;75(4):336-346. doi: 10.1001/jamapsychiatry.2017.4602. PMID 29450462
- [Background] Gujral S, Aizenstein H, Reynolds CF 3rd, Butters MA, Erickson KI. Exercise effects on depression: Possible neural mechanisms. Gen Hosp Psychiatry. 2017 Nov;49:2-10. doi: 10.1016/j.genhosppsych.2017.04.012. PMID 29122145
- [Background] Forteza F, Giorgini G, Raymond F. Neurobiological Processes Induced by Aerobic Exercise through the Endocannabinoidome. Cells. 2021 Apr 17;10(4):938. doi: 10.3390/cells10040938. PMID 33920695
- [Background] Farooq S, Khan T, Zaheer S, Shafique K. Prevalence of anxiety and depressive symptoms and their association with multimorbidity and demographic factors: a community-based, cross-sectional survey in Karachi, Pakistan. BMJ Open. 2019 Nov 19;9(11):e029315. doi: 10.1136/bmjopen-2019-029315. PMID 31748286
- [Background] Diaz-Amaya Y, Star Z, McClure ST. Food security and diet quality, not vitamin D status are significantly associated with depression: Results from NHANES 2015-2018. J Affect Disord. 2024 Feb 15;347:150-155. doi: 10.1016/j.jad.2023.11.071. Epub 2023 Nov 22. PMID 38000464
- [Background] Cipriani A, Furukawa TA, Salanti G, Chaimani A, Atkinson LZ, Ogawa Y, Leucht S, Ruhe HG, Turner EH, Higgins JPT, Egger M, Takeshima N, Hayasaka Y, Imai H, Shinohara K, Tajika A, Ioannidis JPA, Geddes JR. Comparative efficacy and acceptability of 21 antidepressant drugs for the acute treatment of adults with major depressive disorder: a systematic review and network meta-analysis. Lancet. 2018 Apr 7;391(10128):1357-1366. doi: 10.1016/S0140-6736(17)32802-7. Epub 2018 Feb 21. PMID 29477251
- [Background] Bushman, B.A., 2019. Physical activity guidelines for Americans: The relationship between physical activity and health. ACSM's Health & Fitness Journal, 23(3), pp.5-9.
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Brupbacher G, Straus D, Porschke H, Zander-Schellenberg T, Gerber M, von Kanel R, Schmidt-Trucksass A. The acute effects of aerobic exercise on sleep in patients with depression: study protocol for a randomized controlled trial. Trials. 2019 Jun 13;20(1):352. doi: 10.1186/s13063-019-3415-3. PMID 31196147
- [Background] Bennie JA, Teychenne MJ, De Cocker K, Biddle SJH. Associations between aerobic and muscle-strengthening exercise with depressive symptom severity among 17,839 U.S. adults. Prev Med. 2019 Apr;121:121-127. doi: 10.1016/j.ypmed.2019.02.022. Epub 2019 Feb 17. PMID 30786252
- [Background] Edition, F., 2013. Diagnostic and statistical manual of mental disorders. Am Psychiatric Assoc, 21(21), pp.591-643.
- [Background] Alavi NM, Khademalhoseini S, Vakili Z, Assarian F. Effect of vitamin D supplementation on depression in elderly patients: A randomized clinical trial. Clin Nutr. 2019 Oct;38(5):2065-2070. doi: 10.1016/j.clnu.2018.09.011. Epub 2018 Sep 19. PMID 30316534
- [Background] Ait Tayeb AEK, Poinsignon V, Chappell K, Bouligand J, Becquemont L, Verstuyft C. Major Depressive Disorder and Oxidative Stress: A Review of Peripheral and Genetic Biomarkers According to Clinical Characteristics and Disease Stages. Antioxidants (Basel). 2023 Apr 17;12(4):942. doi: 10.3390/antiox12040942. PMID 37107318
- [Background] Ahire, E.D., Keservani, R.K., Balekundri, A., Rajora, A.K. and Surana, K.R., 2024. Effect of nutrients on brain function. In Nutraceutical Fruits and Foods for Neurodegenerative Disorders (pp. 237-248). Academic Press.